CLINICAL TRIAL: NCT01267734
Title: Comparison of the Efficacy and Safety of New Platform Everolimus-eluting Coronary Stent System (Promus Element) With Zotarolimus-eluting Coronary Stent System (Endeavor Resolute) and Triple Anti-platelet Therapy With Double-dose Clopidogrel Anti-platelet Therapy in Patients With Coronary Heart Disease
Brief Title: Harmonizing Optimal Strategy for Treatment of Coronary Artery Stenosis - SAfety & EffectiveneSS of Drug-ElUting Stents & Anti-platelet REgimen
Acronym: HOST-ASSURE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Hyo-Soo Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOST-ASSURE
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Heart Disease
Keywords: Everolimus; Zotarolimus; Cilostazol; Clopidogrel
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EECSS + DDAT (Experimental): Promus Element stent + double-dose clopidogrel anti-platelet therapy
  Interventions: Device: Everolimus-eluting coronary stenting system (EECSS, Promus Element); Drug: Double-dose clopidogrel anti-platelet therapy (DDAT)
- ZECSS + DDAT (Active Comparator): Endeavor Resolute stent + double-dose clopidogrel anti-platelet therapy
  Interventions: Device: Zotarolimus-eluting coronary stenting system (ZECSS, Endeavor Resolute); Drug: Double-dose clopidogrel anti-platelet therapy (DDAT)
- EECSS + TAT (Experimental): Promus Element stent + triple anti-platelet therapy
  Interventions: Device: Everolimus-eluting coronary stenting system (EECSS, Promus Element); Drug: Triple anti-platelet therapy (TAT)
- ZECSS + TAT (Active Comparator): Endeavor Resolute stent + triple anti-platele therapy
  Interventions: Device: Zotarolimus-eluting coronary stenting system (ZECSS, Endeavor Resolute); Drug: Triple anti-platelet therapy (TAT)

INTERVENTIONS:
Device: Everolimus-eluting coronary stenting system (EECSS, Promus Element) — Everolimus-eluting stent
  Other Names: Promus Element
  Arms: EECSS + DDAT; EECSS + TAT
Device: Zotarolimus-eluting coronary stenting system (ZECSS, Endeavor Resolute) — Zotarolimus-eluting stent
  Other Names: Endeavor Resolute
  Arms: ZECSS + DDAT; ZECSS + TAT
Drug: Triple anti-platelet therapy (TAT) — 100mg Aspirin QD + 75mg Clopidogrel QD + 100mg Cilostazol BID for 1 month
  Arms: EECSS + TAT; ZECSS + TAT
Drug: Double-dose clopidogrel anti-platelet therapy (DDAT) — 100mg Aspirin QD + 150mg Clopidogrel QD for 1 month
  Arms: EECSS + DDAT; ZECSS + DDAT

SUMMARY:
Objectives

1. To compare the safety and long-term effectiveness of coronary stenting with the new platform Everolimus-Eluting coronary stenting system (EECSS, Promus Element) compared with the Zotarolimus-Eluting coronary stenting system (ZECSS, Endeavor Resolute) in patients with coronary heart disease (CHD)
2. To determine the short-term efficacy and safety of triple anti-platelet therapy (TAT, Aspirin 100mg qd, Clopidogrel 75mg qd and Cilostazol 100mg bid) compared with double-dose clopidogrel dual anti-platelet therapy (DDAT, Aspirin 100mg qd and Clopidogrel 150mg qd) in patients undergoing percutaneous coronary intervention (PCI) with drug-eluting stents (DES)

Study design Prospective, open-label, 2-by-2 multifactorial, randomized, multicenter trial to test the following in CHD patients

1. Non-inferiority of Promus Element stent compared with Endeavor Resolute stent in reducing target lesion failure (TLF)
2. Non-inferiority of TAT compared with DDAT in reducing net clinical outcome Patients will be randomized in a 2-by-2 factorial manner according to the type of drug eluting stent (EECSS vs. ZECSS) and the type anti-platelet regimen (TAT vs. DDAT). Randomization will also be stratified per presence of DM.

Patient enrollment 3750 patients enrolled at 50 centers in Republic of Korea

Patient follow-up Clinical follow-up will occur at 1, 3, 12, 24, 36 months after the procedure. Angiographical follow-up will be recommended to all participants at 13 months after the procedure. Investigator or designee may conduct follow-up as telephone contacts or office visits.

Primary endpoint

1. Target lesion failure (TLF), defined as a composite of cardiac death, target vessel-related myocardial infarction (MI) and ischemia-driven target lesion revascularization (TLR) up to 12 months for the stent arm
2. Net clinical outcome, defined as a composite of cardiac death, nonfatal MI, CVA and major bleeding by PLATO criteria at 1 month for the anti-platelet arm

DETAILED DESCRIPTION:
Secondary endpoint

1. Clinical and laboratory endpoint at 1 month All death and cardiac death Myocardial infarction (q wave and non-q wave) Stent thrombosis (definite and possible) CVA (hemorrhagic and non-hemorrhagic) Bleeding (major and minor) VerifyNow ASA and VerifyNow P2Y12
2. Clinical endpoint at 12 months All death and cardiac death Target vessel-related MI and all MI (q wave and non-q wave) Target vessel/lesion revascularization (ischemia-driven and all) Stent thrombosis (definite/possible/probable) Net clinical outcome including bleeding (major and minor) Acute success of procedure (device, lesion and procedure)
3. Angiographic (including IVUS or OCT) endpoint at 13 months In-stent & In-segment late loss In-stent & In-segment % diameter stenosis Angiographic pattern of restenosis Neointimal volume, % neointimal volume and % volume obstruction on IVUS or OCT Degree of stent strut endothelialization on OCT

ELIGIBILITY:
General Inclusion Criteria

* Subject must be at least 18 years of age.
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the Promus Element or Endeavor Resolute stents, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have significant lesion (>50% by visual estimate) in any of the coronary arteries, venous or arterial bypass grafts.
* Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia). In subjects with diameter stenosis > 70%, evidence of myocardial ischemia does not have to be documented.

Angiographic Inclusion Criteria

* Target lesion(s) must be located in coronary artery, venous or arterial bypass graft with diameter of ≥ 2.5 mm and ≤ 4.00 mm.
* Target lesion(s) must be amenable for percutaneous coronary intervention.

Exclusion criteria

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Cilostazol, Everolimus, Zotarolimus, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
* Systemic (intravenous) Everolimus or Zotarolimus use within 12 months.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis, known coagulopathy (including heparin-induced thrombocytopenia), abnormal hemogram (Hb<10g/dL or PLT count <100,000/μL) or will refuse blood transfusions
* Patients with severe LV systolic dysfunction (LVEF<25%) or cardiogenic shock
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Symptomatic heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3750 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | 12 months
  Composite of cardiac death, target vessel-related myocardial infarction (MI) and ischemia-driven target lesion revascularization (TLR)
Net clinical outcome | 1 month
  Composite of cardiac death, nonfatal MI, CVA and major bleeding by PLATO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park KW, Kang SH, Kang HJ, Koo BK, Park BE, Cha KS, Rhew JY, Jeon HK, Shin ES, Oh JH, Jeong MH, Kim S, Hwang KK, Yoon JH, Lee SY, Park TH, Moon KW, Kwon HM, Hur SH, Ryu JK, Lee BR, Park YW, Chae IH, Kim HS; HOST-ASSURE Investigators. A randomized comparison of platinum chromium-based everolimus-eluting stents versus cobalt chromium-based Zotarolimus-Eluting stents in all-comers receiving percutaneous coronary intervention: HOST-ASSURE (harmonizing optimal strategy for treatment of coronary artery stenosis-safety & effectiveness of drug-eluting stents & anti-platelet regimen), a randomized, controlled, noninferiority trial. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2805-16. doi: 10.1016/j.jacc.2014.04.013. Epub 2014 May 7. PMID 24814486
- [Derived] Park KW, Kang SH, Park JJ, Yang HM, Kang HJ, Koo BK, Park BE, Cha KS, Rhew JY, Jeon HK, Shin ES, Oh JH, Jeong MH, Kim S, Hwang KK, Yoon JH, Lee SY, Park TH, Moon KW, Kwon HM, Chae IH, Kim HS. Adjunctive cilostazol versus double-dose clopidogrel after drug-eluting stent implantation: the HOST-ASSURE randomized trial (Harmonizing Optimal Strategy for Treatment of Coronary Artery Stenosis-Safety & Effectiveness of Drug-Eluting Stents & Anti-platelet Regimen). JACC Cardiovasc Interv. 2013 Sep;6(9):932-42. doi: 10.1016/j.jcin.2013.04.022. PMID 24050860
- [Derived] Park KW, Park BE, Kang SH, Park JJ, Lee SP, Cha KS, Rhew JY, Jeon HK, Shin ES, Oh JH, Jeong MH, Kim S, Hwang KK, Yoon JH, Lee SY, Park TH, Moon KW, Kwon HM, Chae IH, Kim HS; HOST investigators. The 'Harmonizing Optimal Strategy for Treatment of coronary artery stenosis - sAfety & effectiveneSS of drug-elUting stents & antiplatelet REgimen' (HOST-ASSURE) trial: study protocol for a randomized controlled trial. Trials. 2012 Mar 31;13:29. doi: 10.1186/1745-6215-13-29. PMID 22463698